CLINICAL TRIAL: NCT04485572
Title: Use of Neurodynamic or Orthopedic Tension Tests for the Diagnosis of Lumbar-Sacral and Lumbar Radiculopathies: Study of the Diagnostic Validity
Brief Title: Diagnostic Validity of the Neurodynamic or Orthopedic Tension Tests
Status: Completed | Type: Observational
Sponsor: University of Extremadura (Other)
Collaborators: University of Cadiz (Other)
Responsible Party: Principal Investigator, Elisa María Garrido Ardila, Clinical Professor, University of Extremadura
Other Study IDs: 30/14
Record Dates: First submitted 2020-07-18; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Radiculopathy, Lumbosacral Region
Keywords: Lumbar radiculopathy; Neurodynamic tension tests; Orthopaedic tension tests; Lumbosacral radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Straight Leg Raise test and Bragard test: Patients referred to the radiology department, allocated to undergo MRI scan and neurodynamic tension tests
  Interventions: Diagnostic Test: Straight Leg Raise test (SLR) and Bragard test (B); Diagnostic Test: MRI scan
- Fajersztajn test (F) and Sicard test (S): Patients referred to the radiology department, allocated to undergo MRI scan and neurodynamic tension tests
  Interventions: Diagnostic Test: Fajersztajn test (F) and Sicard test (S); Diagnostic Test: MRI scan
- Passive Neck Flexion test (PNF)and Kernig test (K): Patients referred to the radiology department, allocated to undergo MRI scan and neurodynamic tension tests
  Interventions: Diagnostic Test: Passive Neck Flexion test (PNF)and Kernig test (K); Diagnostic Test: MRI scan
- Slump test (ST) and Dejerine triad (DT): Patients referred to the radiology department, allocated to undergo MRI scan and neurodynamic tension tests
  Interventions: Diagnostic Test: Slump test (ST) and Dejerine triad (DT); Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: Straight Leg Raise test (SLR) and Bragard test (B) — The following neurodynamic and/or orthopedic tension tests were done: the Straight Leg Raise test (SLR), the Bragard test (B) and another test which was the combined test of both (SLR+B)
  Other Names: Index tests
  Groups: Straight Leg Raise test and Bragard test
Diagnostic Test: Fajersztajn test (F) and Sicard test (S) — The following neurodynamic and/or orthopedic tension tests were done: the Fajersztajn test (F), the Sicard test (S) and another test which was the combination of both (F+S)
  Other Names: Index tests
  Groups: Fajersztajn test (F) and Sicard test (S)
Diagnostic Test: Passive Neck Flexion test (PNF)and Kernig test (K) — The following neurodynamic and/or orthopedic tension tests were done: the Passive Neck Flexion test (PNF), the Kernig test (K) and another test which was the combination of both (PNF+K)
  Other Names: Index tests
  Groups: Passive Neck Flexion test (PNF)and Kernig test (K)
Diagnostic Test: Slump test (ST) and Dejerine triad (DT) — The following neurodynamic and/or orthopedic tension tests were done: the Slump test (ST), the Dejerine triad (DT) and another test which was the combination of both (ST+DT)
  Other Names: Index tests
  Groups: Slump test (ST) and Dejerine triad (DT)
Diagnostic Test: MRI scan — All participants will undergo a MRI scan to compare results between the index tests and the Gold Standard
  Other Names: Gold Standard

SUMMARY:
The objective of the present study is to analyse the diagnostic validity of 8 neurodynamic and/or orthopedic tension tests using magnetic resonance imaging as the Gold Standard.

DETAILED DESCRIPTION:
Lumbar radiculopathy is a nerve root disorder which affects quality of life of the patient and it is considered as an important health problem. Therefore, its correct diagnosis is essential. The objective of the present study is to analyse the diagnostic validity of 8 neurodynamic and/or orthopedic tension tests using magnetic resonance imaging as the Gold Standard.

This is an epidemiological study of randomized consecutive cases which was observational, descriptive, transversal, double blinded and followed the STARD (Standards for Reporting Diagnostic accuracy studies) declaration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of lumbar or lumbosacral radiculopathy

Exclusion Criteria:

* Healthy subjects or with a radiculopathy already diagnosed
* subjects with Diabetes, alcoholism, HIV+, herpes zoster infection, cancer, multiple sclerosis, hereditary neuropathy or lumbar surgery
* persons with pacemaker or stent
* known pregnancy
* persons that refused to participate in the study or undergo the MRI scan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population were all the patients referred to the Radiology Department of the 'Puerta del Mar University Hospital' in Cádiz (Spain) to undertake a MRI scan of the lumbar or lumbosacral spine
Sampling Method: Probability Sample
Enrollment: 1887 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the tests | Through study completion, an average of 2 years
  Is is an indicator of the internal validity of the test. The probability that a subject with lumbar or lumbosacral radiculopathy have a positive results in the diagnostic test. It is obtained with the statistical analysis
Specificity of the tests | Through study completion, an average of 2 years
  Is is an indicator of the internal validity of the test. Indicates the percentage of healthy subjects confirmed with a test with negative results. It is obtained with the statistical analysis
Positive and negative predictive values (PV+ and PV-) | Through study completion, an average of 2 years
  Is is an indicator of the internal validity of the test. The range of values are interpreted as: 0-10% null, 10-30% very low; 30-60% low; 60-70% low moderate; 70-80% high moderate; 80-90% high; 90-100% very high.
Likelihood Ratio (LR+ y LR-). | Through study completion, an average of 2 years
  Is is an indicator of the external validity of the test.The range of values and their impact on the clinical utility are: LR+: > 10 great increase, excellent test; 5-10 moderate increase, good test; 2-5: small increase, bad test; < 2: minor increase, useless test. LR-: 0.5-1 minor decrease, useless test; 0,5-0,2 small decrease, bad test; 0,1-0,2 moderate decrease, good test; < 0,1 great decrease, execelent test
Kappa index (K) | Through study completion, an average of 2 years
  It is used to estimate the reliability or accuracy of the tests. The range of values are interpreted as follows: Poor, < 0.20; weak, between 0.21 and 0.40; Moderate, between 0.41 and 0.60; Good, between 0.61 and 0.80; Very good, between 0.80 and 1

IPD SHARING:
Plan to Share IPD: No